CLINICAL TRIAL: NCT05359835
Title: DTPA Chelation for Symptoms After Gadolinium-assisted MRI
Brief Title: DTPA (Diethylenetriaminepenta-acetate) Chelation for Symptoms After Gadolinium-assisted MRI Exposure
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Could not recruit subjects quickly enough
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Lorrin M Koran, MD, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 65231
Record Dates: First submitted 2022-04-26; First posted 2022-05-04 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Gadolinium Deposition Disease
MeSH Terms: interventions — Pentetic Acid

STUDY DESIGN:
Intervention Model Description: Six adult patients aged 18 to 65 who meet diagnostic criteria for Gadolinium Deposition Disease and study inclusion criteria, and are free of exclusion criteria will be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chelation with open-label Ca-DTPA and Zn-DTPA (Experimental): Six chelation treatments utilizing Ca-DTPA on day 1 and Zn-DTPA on day 2. Paired, 2-chelation day treatments will take place at intervals of one week or more.
  Interventions: Drug: Calcium DTPA and Zinc DTPA

INTERVENTIONS:
Drug: Calcium DTPA and Zinc DTPA — Intravenous administration of 2.5 mL (500 mg) of Ca-DTPA over one minute, followed by 900 mL of normal saline infusion over about 90 minutes, followed by 2.5 mL (500 mg) of Ca-DTPA over one minute, followed by infusion of the remaining 100 mL of normal saline over about 10 minutes. Procedure repeated with Zn-DTPA the following day. Two-day procedure repeated at an interval of one week or more for a total of six 2-day treatment sessions.
  Other Names: Diethylenetriaminepenta-acetate

SUMMARY:
The study aims at gathering additional data on the safety and effectiveness of using intravenous administration of the drugs Ca-DTPA/Zn-DTPA to remove the heavy metal gadolinium from the bodies of patients who have retained it and developed symptoms of Gadolinium Deposition Disease following an MRI in which a gadolinium-containing contrast agent was utilized. The outcome data will include measures of symptom relief after as many as six paired Calcium-DTPA/Zinc-DTPA chelation treatments. The study also aims at gathering additional data before and after DTPA treatment regarding levels of certain cytokines in the patients' blood that have been reported to be abnormally elevated in patients with retained gadolinium.

DETAILED DESCRIPTION:
This study aims at gathering additional data on the safety and effectiveness of using intravenous administration of the drug DTPA to remove the heavy metal gadolinium from the bodies of patients who have retained it and developed symptoms of Gadolinium Deposition Disease following an MRI in which a gadolinium-containing contrast agent was utilized. The outcome data will include measures of symptom relief, including chronic pain, skin changes, and cognitive complaints, after as many as six paired Calcium-DTPA/Zinc-DTPA chelation treatments. The study also aims at gathering additional data before and after DTPA treatment regarding levels of certain cytokines (chemical messengers) in the patients' blood that have been reported to be abnormally elevated in patients with retained gadolinium.

DTPA is approved as safe and effective by the federal Food and Drug Administration for the removal of certain radioactive heavy metals, has been in use for more than 60 years, is well tolerated, and has been safely used in three studies, that enrolled 25, 21 and 4 patients respectively who were diagnosed with Gadolinium Deposition Disease.Only the first study reported on symptom improvement, and noted that almost all patients experienced benefit after three paired Calcium-DTPA/Zinc-DTPA chelation treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 - 65 and able to give informed consent.
2. Have had an MRI with contrast at least 3 months and less than 3 years before study enrollment.
3. Have a 24-hour urine analysis 30 days or more post-MRI that documents abnormally high levels of gadolinium excretion.
4. Exhibit within 30 days of the contrast-assisted MRI new onset of 3 or more of the following symptoms:

   1. cognitive disturbance,
   2. extremity pain,
   3. frequent headaches,
   4. chest wall pain,
   5. skin induration,
   6. skin hyper-pigmentation,
   7. skin pain,
   8. arthralgia.
5. Have met these Gadolinium Deposition Disease (GDD) diagnostic criteria for at least 3 months.
6. Received the MRI contrast agent Gadobutrol (Gadovist) and no other MRI contrast agents.

Exclusion Criteria:

1. Diagnosed by the patient's treating MD with an autoimmune or rheumatological disorder such as systemic lupus, rheumatoid arthritis or scleroderma;
2. diagnosed by the patient's treating MD with a condition or conditions that could cause 3 or more of the 8 diagnostic symptoms of GDD;
3. taking a medication or medications that could cause 3 or more of the 8 diagnostic symptoms of GDD;
4. having a condition or conditions and taking a medication or medications that together might account for the presence of 3 or more of the diagnostic symptoms of GDD.
5. Having Wilson's Disease, hemochromatosis, cancer (other than non-melanoma skin cancer), impaired kidney function, or heart disease compromising cardiac function or causing arrhythmia;
6. Participating in another protocol involving a pharmacological or other treatment of GDD.
7. Suffering from a disorder that could raise particular cytokine levels. In addition to autoimmune and rheumatological conditions, these disorders include diabetes mellitus requiring insulin, chronic fatigue syndrome, active infectious disease, covid infection in the past four months, receipt of blood products in the previous 6 months, major depression, and irritable bowel syndrome.
8. Unable for medical reasons or unwilling to discontinue medications known to lower cytokine levels of interest including: lithium, n-acetylcysteine, aspirin, NSAIDs, sertraline and other Selective Serotonin Reuptake Inhibitor antidepressants, and the over-the-counter supplements ashwagandha, astaxanthin, and milk thistle.
9. Prior chelation treatment for GDD.
10. Pregnant, nursing, intending to become pregnant in the next 6 months, unwilling to utilized an approved, effective contraception method during the study's duration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-11 (Estimated); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
0-10 Scale of Pain Severity (Higher is more severe pain) | 2 days before first DTPA treatment
  Rating scale of pain severity
0-10 Scale of Pain Severity | 5-6 days after first 2-day DTPA treatment
  Rating scale of pain severity
0-10 Scale of Pain Severity | 5-6 days after second 2-day DTPA treatment
  Rating scale of pain severity
0-10 Scale of Pain Severity | 5-6 days after third 2-day DTPA treatment
  Rating scale of pain severity
0-10 Scale of Pain Severity | 5-6 days after fourth 2-day DTPA treatment
  Rating scale of pain severity
0-10 Scale of Pain Severity | 5-6 days after fifth 2-day DTPA treatment
  Rating scale of pain severity
0-10 Scale of Pain Severity | 5-6 days after sixth 2-day DTPA treatment
  Rating scale of pain severity
0-10 Scale of Pain Severity | One month after sixth 2-day DTPA treatment
  Rating scale of pain severity

SECONDARY OUTCOMES:
Gadolinium Deposition Disease Symptom rating scale (higher number = symptom is more troubling0 | 2 days before first DTPA treatment treatment
  Scale rating common symptoms seen in Gadolinium Deposition Disease
Gadolinium Deposition Disease Symptom rating scale | 5 to 6 days after first DTPA treatment treatment
  Scale rating common symptoms seen in Gadolinium Deposition Disease
Gadolinium Deposition Disease Symptom rating scale | 5 to 6 days after third DTPA treatment treatment
  Scale rating common symptoms seen in Gadolinium Deposition Disease
Gadolinium Deposition Disease Symptom rating scale | 5 to 6 days after fourth DTPA treatment treatment
  Scale rating common symptoms seen in Gadolinium Deposition Disease
Gadolinium Deposition Disease Symptom rating scale | 5 to 6 days after fifth DTPA treatment treatment
  Scale rating common symptoms seen in Gadolinium Deposition Disease
Gadolinium Deposition Disease Symptom rating scale | 5 to 6 days after sixth DTPA treatment treatment
  Scale rating common symptoms seen in Gadolinium Deposition Disease
Gadolinium Deposition Disease Symptom rating scale | one month after sixth DTPA treatment treatment
  Scale rating common symptoms seen in Gadolinium Deposition Disease
Cognitive Function - Short Form 8a (Promis Item Bank v2.0) (Higher score = more cognitive complaint) | 2 days before first 2-day DTPA chelation
  Measure of cognitive function
Cognitive Function - Short Form 8a (Promis Item Bank v2.0) | 5 to 6 after first 2-day DTPA chelation
  Measure of cognitive function
Cognitive Function - Short Form 8a (Promis Item Bank v2.0) | 5 to 6 after second 2-day DTPA chelation
  Measure of cognitive function
Cognitive Function - Short Form 8a (Promis Item Bank v2.0) | 5 to 6 after third 2-day DTPA chelation
  Measure of cognitive function
Cognitive Function - Short Form 8a (Promis Item Bank v2.0) | 5 to 6 after fourth 2-day DTPA chelation
  Measure of cognitive function
Cognitive Function - Short Form 8a (Promis Item Bank v2.0) | 5 to 6 after fifth 2-day DTPA chelation
  Measure of cognitive function
Cognitive Function - Short Form 8a (Promis Item Bank v2.0) | 5 to 6 after sixth 2-day DTPA chelation
  Measure of cognitive function
Cognitive Function - Short Form 8a (Promis Item Bank v2.0) | one month after sixth 2-day DTPA chelation
  Measure of cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Lorrin M Koran, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Semelka RC, Ramalho M, Jay M, Hickey L, Hickey J. Intravenous Calcium-/Zinc-Diethylene Triamine Penta-Acetic Acid in Patients With Presumed Gadolinium Deposition Disease: A Preliminary Report on 25 Patients. Invest Radiol. 2018 Jun;53(6):373-379. doi: 10.1097/RLI.0000000000000453. PMID 29419708
- [Background] Maecker HT, Wang W, Rosenberg-Hasson Y, Semelka RC, Hickey J, Koran LM. An initial investigation of serum cytokine levels in patients with gadolinium retention. Radiol Bras. 2020 Sep-Oct;53(5):306-313. doi: 10.1590/0100-3984.2019.0075. PMID 33071374
- [Background] Maecker HT, Siebert JC, Rosenberg-Hasson Y, Koran LM, Ramalho M, Semelka RC. Dynamic Serial Cytokine Measurements During Intravenous Ca-DTPA Chelation in Gadolinium Deposition Disease and Gadolinium Storage Condition: A Pilot Study. Invest Radiol. 2022 Jan 1;57(1):71-76. doi: 10.1097/RLI.0000000000000803. PMID 34120127
- [Background] Goetzl EJ, Maecker HT, Rosenberg-Hasson Y, Koran LM. Altered Functional Mitochondrial Protein Levels in Plasma Neuron-Derived Extracellular Vesicles of Patients With Gadolinium Deposition. Front Toxicol. 2022 Jan 12;3:797496. doi: 10.3389/ftox.2021.797496. eCollection 2021. PMID 35295151
- [Background] Denmark D, Ruhoy I, Wittmann B, Ashki H, Koran LM. Altered Plasma Mitochondrial Metabolites in Persistently Symptomatic Individuals after a GBCA-Assisted MRI. Toxics. 2022 Jan 26;10(2):56. doi: 10.3390/toxics10020056. PMID 35202243